CLINICAL TRIAL: NCT00982618
Title: Post Operative Functional Restoration in Patients Undergoing Major Abdominal and Pelvic Laparoscopic Surgery: Effect of Perioperative Intravenous Lidocaine
Brief Title: Functional Restoration After Abdominal and Pelvic Laparoscopic Surgery: Effect of Perioperative Intravenous Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Gabriele Baldini, Assistant Professor, Dr, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEN-06-023
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Colon Cancer; Inflammatory Bowel Diseases; Diverticulitis
MeSH Terms: conditions — Colonic Neoplasms; Inflammatory Bowel Diseases; Diverticulitis | interventions — Lidocaine; Anesthesia, Epidural; Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LIDOCAINE group (Experimental): LIDOCAINE group : Beside general anesthesia, patients will receive intravenous lidocaine bolus 1.5 mg/kg just prior induction and an infusion of lidocaine 2mg/kg/h will be started and maintained during the whole surgical procedure. Entering the recovery room, this infusion will be decreased at the rate of 1mg/kg/hour for the 48 first hours
  Interventions: Drug: Lidocaine
- Epidural Group (Experimental): Epidural Group: Beside general anesthesia, patient will receive epidural freezing medication for 48 hours.
  Interventions: Procedure: Epidural Block
- PCA group (Active Comparator): Beside general anesthesia, the patients will receive neither lidocaine nor epidural catheter. The patients will receive the same analgesia protocol consisting of PCA morphine for a total duration of 48 hours.
  Interventions: Drug: PCA Morphine

INTERVENTIONS:
Drug: Lidocaine — 1% Lidocaine 1mg/kg/hr IV drip x 48hr
  Other Names: Intravenous local anesthetic infusion
  Arms: LIDOCAINE group
Procedure: Epidural Block — 0.1% Epidural bupivacaine + Morphine 0.02 mg/ml drip via epidural x48 hr
  Other Names: Thoracic epidural analgesia
  Arms: Epidural Group
Drug: PCA Morphine — PCA Morphine is set to the patient for 48 hours postoperative. 2 mg. of morphine is given to a patient as much as patient requires, maximum at every 7 minutes.
  Other Names: Patient Control Analgesia Morphine.
  Arms: PCA group

SUMMARY:
This is a blinded randomized controlled trial in patients undergoing laparoscopic colon surgery. The aim of this study is to assess whether perioperative intravenous lidocaine has an impact on the early post operative physical activity recovery of patients scheduled for laparoscopic colon surgery.

Twenty patients will receive thoracic epidural analgesia, twenty patients will receive intravenous lidocaine plus patient-controlled analgesia (PCA) and twenty patients will receive only PCA.

Hypothesis: patients receiving perioperative intravenous lidocaine, post operative recovery will be faster and decrease pain intensity, opioid consumption and side effects, length of hospital stay; probably as a result of a significant opioid sparing and attenuated inflammatory response.

DETAILED DESCRIPTION:
This is a blinded randomised study of patients undergoing major laparoscopic abdominal and pelvic surgery. The first group of patients will receive thoracic epidural analgesia, the second group will receive perioperative intravenous lidocaine, the third group will PCA alone and the last group will receive spinal analgesia. Functional restoration assessed by self-administered quality of Life questionnaires (SF-36, CHAMPS, ICFS) and 2 and 6 min walking test will be assessed in the two groups at 3 and 8 weeks after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo laparoscopic colonic resection

Exclusion Criteria:

* patients who have trouble to understand, read or communicate either in French or in English
* dementia
* patients suffering from severe physical disability (arthritis, neuromuscular dysfunction, stroke, paraplegia) or inability to walk or conduct daily activity
* patients suffering from severe cardiac or respiratory disease (status ASA IV)
* patients suffering from metastatic carcinoma
* patients who have a history of chemoradiation within the six months preceding surgery
* allergy to lidocaine
* morbid obesity

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Postoperative functional recovery | daily during hospitalization, and at 4 and 8 weeks after the surgery

SECONDARY OUTCOMES:
postoperative pain | daily during hospitalization
opioid consumption | daily during hospitalization
opioid side effects | daily during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, Professor, Principal Investigator — McGill University Healt Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada